CLINICAL TRIAL: NCT03341104
Title: Evaluation of Intraoperative, Local Site Injections of Liposomal Bupivacaine as an Alternative to Standard Local Anesthetics in Patients Undergoing Total Hip Arthroplasty
Brief Title: Evaluation of LB in THA
Status: Completed | Type: Observational
Sponsor: OSF Healthcare System (Other)
Collaborators: University of Illinois College of Medicine at Peoria (Other)
Responsible Party: Principal Investigator, Ed Rainville, Clinical Pharmacy Supervisor, OSF Healthcare System
Other Study IDs: hipstudy2017
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Hip Disease
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bupivacaine liposome — Replace bupivacaine with bupivacaine liposome
  Other Names: bupivacaine

SUMMARY:
This study aims to compare the effectiveness of liposomal bupivacaine (LB) versus standard of practice local injection containing plain bupivacaine.

DETAILED DESCRIPTION:
Investigation of liposomal bupivacaine to determine if this drug is a valid alternative to standard of care local anesthesia based on evaluation in total hip arthroplasty This is a retrospective cohort study of consecutive patients undergoing THA at 3 hospitals within a U.S. healthcare system from January 2013 to July 2016. The control group received the standard of care undergoing THA (plain bupivacaine or ropivacaine), while the LB group received a mixture containing this drug as the alternative to the standard care. The outcome variables include hospital length of stay, readmissions, total hospital costs, patient pain scores, discharge disposition, morphine equivalent opioid consumption, and postoperative patient ambulation. Generalized linear models were employed to examine aforementioned outcomes controlling for age, gender, race, BMI, alcohol use, tobacco use, and surgeons..

ELIGIBILITY:
Inclusion Criteria:

* Males or females over the age of 18
* have undergone a THA surgery during the period of interest January 2013 to July 2016).

Exclusion Criteria:

* excluded from the study based on the following criteria:

  1. Concurrent, painful, physical condition or concurrent surgery that may require analgesic treatment in the postoperative period for pain that is not strictly related to the surgical treatment;
  2. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder; and
  3. Significant renal or hepatic insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to acute care facilities for total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Comparing physical function of the control group with the experimental group | 43 months
  distance in feet walked
Comparing length of stay in acute care facility of the control group with the experimental group | 43 months
  number of days
Comparing total hospital costs of the control group with the experimental group | 43 months
  Number of dollars

CONTACTS AND LOCATIONS:
Overall Officials: Ed Rainville, Principal Investigator — OSF HealthCare Ssytem

IPD SHARING:
Plan to Share IPD: No